CLINICAL TRIAL: NCT03471611
Title: A Phase 1, Feasibility Study Testing the Safety and Feasibility of Intracoronary CD34+ Cell Administration on Coronary Endothelial Function in Patients With Early Coronary Atherosclerosis
Brief Title: Study of Intracoronary CD34+ Cell Administration in Patients With Early Coronary Atherosclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-005743
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Atherosclerosis, Coronary
MeSH Terms: conditions — Coronary Artery Disease | interventions — betibeglogene autotemcel; Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with Endothelial Dysfunction (Experimental): Subjects will be treated with Granulocyte Colony-Stimulating Factor (G-CSF) for 5 days at a dose of 5 mg/kg twice daily. When count of CD34+ cells is sufficient, the CD34+ cells will be collected by apheresis. Autologous CD34+ cells will be injected into the subjects at a rate of 10 ml/min.
  Interventions: Drug: Autologous CD34+ Cells; Drug: Granulocyte Colony-Stimulating Factor (G-CSF)

INTERVENTIONS:
Drug: Autologous CD34+ Cells — The dose will be 1x10^5 cells/kg, injected at the rate of 10 ml/min
Drug: Granulocyte Colony-Stimulating Factor (G-CSF) — 5mg/kg twice daily
  Other Names: Neupogen; Neulasta

SUMMARY:
How safe and effective are CD34+ cell intracoronary injections for treating coronary endothelial dysfunction (CED)?

DETAILED DESCRIPTION:
This is an open label, phase I study to determine safety and efficacy of CD34+ cells in the treatment and management of CED and early atherosclerosis. Coronary endothelial function will be assessed in all patients by the administration of intracoronary acetylcholine. Patients with endothelial dysfunction who meet study inclusion criteria will receive granulocyte cell stimulating factor (G-CSF), followed by apheresis. The mobilized peripheral cell product will be processed for selection of CD34+ stem cells, and the purified CD34+ cells will be administered intracoronary during cardiac catheterization. The patients will undergo repeat endothelial function assessment 6 months post-procedure, as well as clinical assessments as described below either via in-person assessment by a nurse or physician, or via phone-call using a standardized questionnaire at 1, 3, and 6 month follow-up visits. At one month, the patient will undergo basic laboratory testing including troponin levels, complete blood count (CBC), electrolyte panel, liver function testing and ECG. At 3 months, the patients will receive a phone follow-up by the study coordinator who will assess the patient for any clinical deterioration or significant worsening in symptoms. At 6 months, the patients will return for a clinical visit, which will include physical examination, basic laboratory testing and follow-up acetylcholine study with angiography to assess for change in endothelial function. The first three patients will be sequentially enrolled, and subsequent enrollment will be held until one month follow-up. Provided there are no safety concerns at this time, enrollment will continue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of coronary endothelial dysfunction based on coronary angiogram and acetylcholine comprehensive coronary physiology study
* Able to provide informed written consent and willing to participate in all required study follow-up assessments

Exclusion Criteria:

* Acute coronary syndrome or continuous/ongoing chest pain - unremitting and unresponsive to nitroglycerin or rest - persisting 4 or more days before stent placement. If the chest pain syndrome is transient and/or intermittent - even if it began more than 3 days prior to admission - the patient is not excluded.
* Subjects in cardiogenic shock (systolic pressure < 80mm/Hg, on vasopressors or intraaortic counter pulsation) at the time of consenting. Subjects who recover from cardiogenic shock by the time of consenting are eligible.
* Subjects unable to receive antiplatelet agents (e.g. aspirin, clopidogrel, ticlopidine,prasugrel, etc).
* Abnormal laboratory values (Hgb <11 mg/dL; glomerular filtration rate (GFR)<50; liver function tests (LFTs)>2x upper limit of normal).
* Subjects receiving warfarin who have an international normalized ratio (INR) >2 at the end of the screening phase or with major bleeding requiring active transfusion support.
* Subjects with severe cardiac valvular disease expected to undergo surgery within 1 year.
* Subjects with known severe immunodeficiency states (AIDS).
* Significant coronary artery disease on coronary angiogram
* Cirrhosis requiring active medical management.
* Malignancy requiring active treatment (except basal cell skin cancer).
* Subjects with documented active alcohol and /or other substance abuse.
* Females of child bearing potential unless a pregnancy test is negative within 7 days of the bone marrow harvest.
* Re-occlusion of the infarct related artery (IRA) prior to the infusion procedure.
* Planned revascularization intervention during the next 6 months. (A second PCI can be performed if done prior to qualifying cardiovascular magnetic resonance imaging (CMR) at least 96 hours post primary PCI).
* Participation in an ongoing investigational trial.
* Active or suspected bacterial infection requiring systemic intravenous antibiotics.
* Additional factors deemed unsuitable for trial enrollment per discretion of principal investigator
* Inmates

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events | 12 months
Number of subjects experiencing serious adverse events | 12 months
Number of subjects experiencing Major Adverse Cardiovascular Events (MACE) | 12 months
  The most commonly reported major cardiovascular adverse events (MACE) include myocardial infarction, heart failure, percutaneous cardiac intervention, coronary artery bypass grafting, malignant dysrhythmia, cardiac shock, implantable cardiac defibrillator, malignant dysrhythmia and death.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Corban MT, Toya T, Albers D, Sebaali F, Lewis BR, Bois J, Gulati R, Prasad A, Best PJM, Bell MR, Rihal CS, Prasad M, Ahmad A, Lerman LO, Solseth ML, Winters JL, Dietz AB, Lerman A. IMPROvE-CED Trial: Intracoronary Autologous CD34+ Cell Therapy for Treatment of Coronary Endothelial Dysfunction in Patients With Angina and Nonobstructive Coronary Arteries. Circ Res. 2022 Feb 4;130(3):326-338. doi: 10.1161/CIRCRESAHA.121.319644. Epub 2021 Dec 20. PMID 34923853
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials